CLINICAL TRIAL: NCT06671067
Title: Noninvasive Assessment of Pulmonary Fluid Levels by Remote Dielectric Sensing (ReDS™) Technology to Improve Cardiac Insufficiency During Ischemia-reperfusion and Clinical Outcomes in Myocardial Infarction
Brief Title: Noninvasive Assessment of Pulmonary Fluid Levels by Remote Dielectric Sensing Technology to Improve Cardiac InsUfficieney During Ischemia-Reperfusion and Clinical Outcomes in MyocArdiaL Infarction
Acronym: NATURAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Chief Physician, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NATURAL
Record Dates: First submitted 2024-10-29; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Acute Myocardial Infarction; Acute Decompensated Heart Failure (ADHF)
Keywords: Remote dielectric sensing system; Acute myocardial infarction; Acute heart failure; Clinical outcomes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Routine care group (No Intervention): AMI patients with cardiac insufficiency following coronary revascularization who receive the routine care without ReDS guiding
- ReDS-guided care group (Experimental): AMI patients with cardiac insufficiency following coronary revascularization who receive the ReDS guiding care
  Interventions: Device: Remote dielectric sensing system

INTERVENTIONS:
Device: Remote dielectric sensing system — The remote dielectric sensing (ReDS) system is a non-invasive medical device that emits a low-power electromagnetic signal through the chest and lungs, which can accurately measure changes in lung fluid concentration.
  Arms: ReDS-guided care group

SUMMARY:
To explore whether a ReDS-guided strategy for AMI patients with cardiac insufficiency following coronary flow reperfusion is superior to routine care for improving outcomes.

DETAILED DESCRIPTION:
The remote dielectric sensing (ReDS) system is a non-invasive medical device that emits a low-power electromagnetic signal through the chest and lungs, which can accurately measure changes in lung fluid concentration. Previous studies suggest that ReDS-guided management may have the potential role in the diagnosis and treatment of acute heart failure (AHF): (1) Assessment of real-time volume status: Patients with AHF are often accompanied by volume overload, especially pulmonary congestion, which is one of the main risk factors for readmission; (2) Establishment of treatment strategy: The ReDS-SAFE HF study showed that the AHF treatment strategy based on the ReDS measurement could significantly reduce the readmission rate and the clinical outcomes after discharge; (3) Determine time to discharge: The study ReDS-SAFE HF also suggests ReDS measurement can aid physicians to determine the appropriate time to discharge by monitoring changes in the volume of lung fluid, which can relatively avoid the risk of early or late discharge.

Acute myocardial stunning and injury combined with cardiac insufficiency is one common complication of acute myocardial infarction (AMI), the large infarcted area of the left ventricular anterior wall can lead to heart pump failure, which will cause pulmonary edema and acute decompensated heart failure (ADHF) in the long-term recovery. Although cardiomyocytes do not completely lose their activity following the cardiac circulatory reperfusion, it still requires a long period for the myocardium to restore normal function, which closely related to the basal myocardial status, number of coronary lesions, area of myocardial infarction, and time of reperfusion. Long-time loss of myocardial activity then results in irreversible myocardial remodeling of patients in and seriously impacts the life quality of life of AMI patients. Therefore, it is particularly important to find an effective convenient management scheme to improve cardiac insufficiency following ischemic reperfusion in AMI patients. Among these patients, acute ischemic myocardium and cardiac dysfunction could simultaneously induce rapid adaptive alterations in lung fluid, which provides an indicative parameter in the clinical and could be well-determined by the ReDS devices.

This study sought to explore whether a ReDS-guided strategy for AMI patients with cardiac insufficiency following coronary flow reperfusion is superior to routine care for improving outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were required to be aged ≥ 18 years and to be hospitalized for a primary diagnosis of AMI,
2. AMI patients accompanied by cardiac insufficiency following coronary revascularization, which is characterized by the symptoms and signs of fluid overload, regardless of left ventricular ejection fraction (LVEF), and have an N-terminal pro-B-type natriuretic peptide (NT-proBNP) concentration of ≥ 400 pg/L or a BNP concentration of ≥ 100 pg/L.

Exclusion Criteria:

1. Patient's physical characteristics that prevented the use of the ReDS system (height of <155 or >190 cm; body mass index of <22 or >39 kg/m2)
2. Patients with chronic obstructive pulmonary disease or other lung diseases that might confound ReDS values
3. Patients with a left ventricular assist device or undergoing cardiac transplantation;
4. Patients with congenital heart malformations or intrathoracic mass that would affect right lung anatomy;
5. Patients with end-stage renal disease on hemodialysis;
6. Patients whose life expectancy less than 12 months due to noncardiac comorbidities
7. Patients who participate in another randomized studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac event (MACE) | 1 year
  The primary outcome is the MACE that is defined as a composite of all-cause death and HF readmission.

SECONDARY OUTCOMES:
All-cause death | 1 year
HF readmission | 1 year
  HF readmission was defined as a minimum of an overnight hospitalization for a patient presenting with symptoms and signs of HF or requiring intravenous diuretics
The length of hospital readmission stay | 30 days
  The length of hospital readmission stay
Quality of life (QOL) | 1 year
  The quality of life was assessed according to Minnesota Living with Heart Failure Questionnaire (MLHFQ). The 21 items of MLHFQ are rated on six-point Likert scales, representing different degrees of impact of HF on patient's QOL, from 0 (no) to 5 (very much). It provides a total score (range 0-105), from best to worst QOL.

OTHER OUTCOMES:
Changes in BNP levels | 30 days
  Changes in BNP levels
Changes in NYHA functional class | 30 days
  Changes in NYHA functional class

CONTACTS AND LOCATIONS:
Overall Officials: Yidong Wei, M.D., Ph.D., Principal Investigator — Shanghai 10th People's Hospital
Locations (6):
- China (6):
  - Huaihe Hospital of Henan University, Kaifeng, Henan
  - Kaifeng Central Hospital, Kaifeng, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Seventh People's Hospital of Shanghai University of Traditional Chinese Medicine Shanghai, Shanghai, Shanghai Municipality
  - Songjiang Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided